CLINICAL TRIAL: NCT00213707
Title: Liver Transplanted Patients for HCV Related End Stage Liver Disease.Functional Role of Blood Circulating Dendritic Cells in the Pathogenesis of Hepatitis C Virus Infection During Liver Transplantation.
Brief Title: Study of the Role of Dendritic Cells in the Recurrence of Hepatitis C After Liver Transplantation. Analysis of Hepatitis C Virus (HCV) Quasispecies Evolution.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Other Study IDs: 2864
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: HCV Infection
Keywords: Dendritic cells; liver transplantation; hepatitis C virus; quasispecies; virological markers; biochemical markers; immunological markers; clinical markers
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Re-infection of the liver graft occurs universally following liver transplantation for HCV-induced end stage liver disease. Interestingly, the manifestation of HCV infection ranging from an asymptomatic carrier state to rapid progression to liver cirrhosis is extremely variable from one patient to another. The host and viral factors being responsible for the different course of HCV infection are poorly understood. Our study will focus on dendritic cells which are known to play a critical role in the control of viral infection. Viral factors (quasispecies evolution) will also be analysed and Th1 Th2 cytokines produced in the serum evaluated.Thirty liver transplanted patients will be included : 20 patients transplanted for HCV-related disease and 10 controls transplanted for non HCV-related disease. Blood samples will be taken just before transplantation and at different time -points up to 5 years after transplantation. Function of blood monocyte-derived DC will be evaluated. Circulating blood plasmacytoid (pDC) and myeloid DC (mDC) sub-populations will be enumerated. HCV quasispecies evolution will be analysed. This study may help to define prognostic markers on progression of hepatitis C in liver transplantation and allow the development of new immunotherapeutic drugs

ELIGIBILITY:
Inclusion Criteria:

Liver transplanted HCV infected patients :

* Adults, HIV(-),HBV(-)
* liver transplanted for an end stage liver disease associated to HCV.
* Genotype determined
* written agreement to participate to the study

Control patients :

* Adults, HIV(-), HBV(-), HCV(-)
* liver transplanted for a non HCV liver disease
* written agreement to participate to the study.

Exclusion Criteria:

* HIV(+), HBV(+)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for liver transplantation indicated after chronic hepatitis C.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2003-05; Primary Completion 2010-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Function of blood circulating DC at day 7 and 1, 3, 6, 9, 12 months, 2 and 5 years after liver transplantation depending on the clinical outcome (mild or severe hepatitis, cirrhosis). | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Stoll-Keller, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (1):
- Francoise Stoll-Keller, Strasbourg, France